CLINICAL TRIAL: NCT05710627
Title: Evaluation of Percutaneous Tenotomy of the Gluteus Medius and Iliotibial Band for Greater Trochanteric Pain Syndrome (GTPS): A Randomized Clinical Trial
Brief Title: Evaluation of TENEX for Greater Trochanteric Pain Syndrome (GTPS)
Acronym: RCT GTPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-14588
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Greater Trochanteric Pain Syndrome

STUDY DESIGN:
Intervention Model Description: 100 patients will be enrolled in the TENEX group and 50 patients in the control group accounting for 10% rate of loss-to-follow-up. 10 pre computer-generated blocks, consisting of 15 patients in each block, will be generated. In each block, 5 patients will be assigned to CMM and 10 to the Tenex group. Patients will be assigned to each group by the order that computer has created.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): Standard of care
- Treatment (Experimental): TENEX device will be used
  Interventions: Device: TENEX

INTERVENTIONS:
Device: TENEX — Use of TENEX device for sectioning of the gluteus medius and ITB tendons.
  Arms: Treatment

SUMMARY:
The objective of this study is to evaluate how an ultrasound-guided percutaneous procedure, TENEX, can help people with chronic hip pain resulting from a condition called Greater Trochanteric Pain Syndrome (GTPS) and to characterize the efficacy of percutaneous tenotomy (PUT) using TENEX®, a device used for the treatment of various tendinopathies. In this study an ultrasound (US) is performed to guide the partial release of gluteus medius and minimus and Iliotibial band tendons in patients diagnosed with refractory Greater Trochanteric Pain Syndrome (GTPS) vs control. The investigator team hypothesizes that the new TENEX can improve the pain level for individuals with GTPS to help those individuals perform their activities of daily living (ADLs), e.g., walking, standing, and side-lying, as well as demonstrate less medication utilization. The study predicts that this percutaneous outpatient procedure can decrease pain, increase mobility, and decrease medication utilization.

The study team hypothesizes that PUT can improve the pain level and function for individuals suffering with GTPS. The study will assess walking, standing, and side-lying tolerance, as well as medication utilization. The investigator team predicts that this percutaneous outpatient procedure can decrease pain and medication utilization while increasing mobility.

DETAILED DESCRIPTION:
Greater trochanteric pain syndrome (GTPS) is one of the most common causes of lateral hip pain in adults. GTPS is repetitive overload tendinopathy of the gluteus medius (GMed) and Iliotibial band (ITB), which play a primary role in hip abduction and pelvic stabilization in walking, stair climbing, running and standing on one leg. It is thought that the core pathology is greater trochanteric bursitis (TB) with or without coexisting gluteal tendinopathy. Some common etiologies include prolonged excessive pressure to the area, injury to the side of the hip, and repetitive movements; however, local steroid injections to the greater TB are not often successful over the long-term. The best estimates of prevalence are from a large, community-based study with over 3000 adults aged 50 to 70 years, in which unilateral GTPS was present in 15 percent of women and 6.6 percent of men. Patients who have not improved after at least 12 months of conservative medical management (CMM), including physical therapy, oral medications, or a local steroid injection have no other conservative treatment recourse. Open surgery for GMed or ITB tears is not recommended unless a tear is diagnosed on MRI. Based on a published study, a 60% improvement was shown in pain with the performance of TENEX of the GMed.

The purpose of this project is to study the outcome of GMed and ITB PUT on CMM refractory GTPS. We want to quantify and show the scales of the pain in pre-operative and post-treatment cases. We also want to see how effective the surgery is in specific terms of pain levels because GTPS is a pain syndrome and reduction in pain level is the most important clinical factor.

Patient Reported Outcome Measure (PROM) is one of the main outcomes that medical research is validated with and through this study we want to show the most important outcome of GTPS i.e., pain level (PROM for GTPS). Previous studies which focused on surgical outcomes have been mostly single-center trials.

Pain and mobility impact patients' Quality of Life (QoL) and medical cost burden due to unemployment, psychosocial well-being, and functional dependence. The standard of care offered to address the pain and mobility needs of those with GTPS is to provide CMM, followed by open or arthroscopic surgery if surgery is indicated. However, there is a treatment gap for those patients who have failed CMM and are not surgical candidates. The authors submit that TENEX of the GMed and ITB may address this gap. The results from this research may have broad impacts on the treatment algorithm for patients with GTPS.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-90
* People with GTPS of all different levels and etiologies confirmed with MRI or CT scan
* Ability to give informed consent forms independently
* Failed conservative medical treatment for at least 6 months

Exclusion Criteria:

* Significant mobility restrictions; people using wheelchairs
* Pregnancy
* Previous surgery to the GMed or ITB

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-03-11 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Pain Level | Baseline (before treatment), 1 month, 3 months, 6 months, 1 year, and 2 years
  The difference in pain levels in patients before and after the procedure. Pain levels (NRS scale) recorded in the pre-operative visit will be compared to the pain levels at follow-up (FU) visits. The Numeric rating scale (NRS) is a pain screening tool used to assess pain severity using a 0-10 scale, with 0 meaning no pain and 10 meaning the worst pain imaginable. Pain level scores will be summarized by study arm. Achievement of 50% reduction in pain level from baseline at 6 months post treatment will be considered successful.

SECONDARY OUTCOMES:
Quality of Life using the European Quality of Life 5 Dimensions 5 Level Version (EQ-5D-5L) | Baseline (before treatment), 1 month, 3 months, 6 months, 1 year, and 2 years
  A comparative analysis between TENEX to conventional medical treatments will be conducted using the EQ-5D-5L. Walking, side-lying, sit-to-stand transfers, and medication utilization will be assessed. The EQ-5D-5L is a descriptive system which comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1- digit number that expresses the level selected for that dimension. The digits for the five dimensions are combined into a five-digit number that describes the patient's health state. Results will be summarized by study arm.

CONTACTS AND LOCATIONS:
Overall Officials: Sayed E. Wahezi, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Segal NA, Felson DT, Torner JC, Zhu Y, Curtis JR, Niu J, Nevitt MC; Multicenter Osteoarthritis Study Group. Greater trochanteric pain syndrome: epidemiology and associated factors. Arch Phys Med Rehabil. 2007 Aug;88(8):988-92. doi: 10.1016/j.apmr.2007.04.014. PMID 17678660
- [Background] Baker CL Jr, Mahoney JR. Ultrasound-Guided Percutaneous Tenotomy for Gluteal Tendinopathy. Orthop J Sports Med. 2020 Mar 19;8(3):2325967120907868. doi: 10.1177/2325967120907868. eCollection 2020 Mar. PMID 32232066
- [Background] Del Buono A, Papalia R, Khanduja V, Denaro V, Maffulli N. Management of the greater trochanteric pain syndrome: a systematic review. Br Med Bull. 2012 Jun;102:115-31. doi: 10.1093/bmb/ldr038. Epub 2011 Sep 4. PMID 21893483
- [Background] Mellor R, Grimaldi A, Wajswelner H, Hodges P, Abbott JH, Bennell K, Vicenzino B. Exercise and load modification versus corticosteroid injection versus 'wait and see' for persistent gluteus medius/minimus tendinopathy (the LEAP trial): a protocol for a randomised clinical trial. BMC Musculoskelet Disord. 2016 Apr 30;17:196. doi: 10.1186/s12891-016-1043-6. PMID 27139495
- [Background] Chandrasekaran S, Lodhia P, Gui C, Vemula SP, Martin TJ, Domb BG. Outcomes of Open Versus Endoscopic Repair of Abductor Muscle Tears of the Hip: A Systematic Review. Arthroscopy. 2015 Oct;31(10):2057-67.e2. doi: 10.1016/j.arthro.2015.03.042. Epub 2015 May 29. PMID 26033462
- [Background] Wahezi SE, Patel A, Yerra S, Naeimi T, Sayed D, Oakes D, Ortiz N, Yee M, Yih C, Sitapara K, Schulz J, Kohan L, Rosenburg J, Schwechter E, Chan F, Gonzalez D, Baker C. Percutaneous Ultrasound-Guided Tenotomy of the Iliotibial Band for Trochanteric Pain Syndrome: A Longitudinal Observational Study With One-Year Durability Results. Pain Physician. 2023 Jul;26(4):393-401. PMID 37535779